CLINICAL TRIAL: NCT07122440
Title: Évaluation Des Facteurs Pronostiques et de l'évolution Des mastoïdites aigües Dans la région Grand-Est
Brief Title: Outcomes and Prognostic Factors of Acute Mastoiditis in the Grand-Est Region
Acronym: MAGE
Status: Completed | Type: Observational
Sponsor: Cécile RUMEAU (Other)
Responsible Party: Sponsor-Investigator, Cécile RUMEAU, Head of Otolaryngology, Central Hospital, Nancy, France
Organization: Central Hospital, Nancy, France (Other)
Other Study IDs: 2023PI213
Record Dates: First submitted 2024-01-03; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Acute Mastoiditis
Keywords: acute mastoiditis; prognostic; mastoiditis complications

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: acute mastoiditis — retrospective data collection from clinical charts

SUMMARY:
There is an increased incidence of acute mastoïditis and a lack of homogeneity in management. The investigator aim to refine the epidemiological knowledge on this pathology.

Data of children with acute mastoiditis of the last ten years in five hospitals of the North-East of France (University Hospitals of Nancy, Strasbourg, Dijon, Besançon and the Regional Hospital of Metz-Thionville) will be analyzed.

DETAILED DESCRIPTION:
Acute mastoiditis is a bacterial infection of the middle ear cavities, associated with destructive damage of the mastoid bone, complicating acute otitis media. It affects infants and young children and its complications can be serious, including neurological sequelae.

These complications can be divided into two categories according to their topography:

* intracranial complications : thrombophlebitis, meningitis, epidural abscess, and cerebral empyema.
* Extracranial complications subperiosteal abscess, Bezold's abscess, peripheral facial paralysis, labyrinthitis, and temporomandibular joint arthritis.

Incidence ranges from 1.2 to 6 per 100,000 children per year, with a trend of increasing cases with the increase in the proportion of Fusobacterium Necrophorum infections, described as frequent provider of complications. This observation is shared by the ENT practitioners of the CHRU of Nancy.

The management of mastoiditis is medico-surgical, but the therapeutic algorithms vary according to the centers and countries. The exact place of surgery is discussed in uncomplicated cases, despite recent meta-analyses. In France, no therapeutic algorithm is currently proposed by ENT societies.

Given this double observation of increased incidence and lack of homogeneity in the management of mastoiditis, it appears to be useful to refine the epidemiological knowledge on this pathology.

Therefore, we will analyze data of children with acute mastoiditis of the last ten years in five hospitals of the North-East of France : University Hospitals of Nancy, Strasbourg, Dijon, Besançon and the Regional Hospital of Metz-Thionville.

ELIGIBILITY:
Inclusion Criteria:

* All patients under 15 years of age
* Supported in one of the ENT or pediatric services of the four investigation centers
* Between January 1, 2014 and July 31, 2024
* With a diagnosis of acute mastoiditis

Exclusion Criteria:

* Patient with history of cholesteatoma or cochlear implantation

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Cf Eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 326 (Actual)
Dates: Start 2024-03-02 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Prognostic factors of recovery in children hospitalized for mastoiditis in the region Grand-Est of France between 2014 and 2024 | From January 2014 to July 2024
  The primary outcome was recovery by Day 5, i.e., recovery on the fifth day of hospitalization.
  Recovery was a composite outcome based on three subcriteria:
  * (i) absence of fever (body temperature ≥ 38°C);
  * AND (ii) absence of neutrophilia (neutrophil count > 8.5 G/L);
  * AND (iii) absence of local symptoms (i.e., otalgia or ear inflammation).
  Patients presenting with fever OR neutrophilia OR local clinical symptoms on Day 5 or later were classified as not recovered by Day 5. Fever and local symptoms are monitored by the nursing staff several times a day during the hospitalization. The neutrophil count is measured as part of the laboratory test, performed on the day of hospital admission, and carried out multiple times during hospitalizations. The absence of follow-up laboratory testing suggests clinical improvement.
  The abovementioned outcomes were extracted, as well as variables known or suspected to be associated with mastoiditis recovery or complications.

SECONDARY OUTCOMES:
Evolution of complication rate of mastoiditis between January 2014 and July 2024 | From January 2014 to July 2024
  Intracranial complications were defined by the presence of thrombophlebitis, meningitis, epidural abscess, and cerebral empyema.
  Extracranial complications included subperiosteal abscess, Bezold's abscess, peripheral facial paralysis, labyrinthitis, and temporomandibular joint arthritis.
Factors associated with complicated acute mastoïditis | From January 2014 to July 2024
  Intracranial complications were defined by the presence of thrombophlebitis, meningitis, epidural abscess, and cerebral empyema.
  Extracranial complications included subperiosteal abscess, Bezold's abscess, peripheral facial paralysis, labyrinthitis, and temporomandibular joint arthritis.
  The abovementioned outcomes were extracted, as well as variables known or suspected to be associated with mastoiditis recovery or complications. These variables were patients' demographic characteristics (age, gender, hospital center), medical history (prematurity, surgery), pre-hospital care (delay between symptom onset and hospitalization, antibiotic treatment before admission), medical care during the hospitalization (surgery, anti-inflammatory treatment, empirical and targeted antibiotic therapy), biological results (date of laboratory tests, C-reactive protein, leucocytes, neutrophils), bacteriological results (date and type of specimen, bacteria identified).

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Center of Nancy, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No